CLINICAL TRIAL: NCT02675088
Title: Randomized Phase III Study Comparing Different Thoracic Radiotherapy Regimens in Patients With Extensive Stage Small Cell Lung Cancer Who Respond to Chemotherapy
Brief Title: Comparable Study of Different Thoracic Radiotherapy Regimens for Extensive Stage Small Cell Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Sun Yat-sen University (Other); Fudan University (Other); West China Hospital (Other); Zhejiang Cancer Hospital (Other); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Luhua Wang, Vice President of Cancer hospital of CAMS, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-L-045/1
Record Dates: First submitted 2016-02-03; First posted 2016-02-05 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Carcinoma, Small Cell; Lung Neoplasms
Keywords: Extensive Stage Small Cell Lung Cancer; thoracic radiotherapy; radiotherapy regimen
MeSH Terms: conditions — Carcinoma, Small Cell; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- high-dose TRT (Experimental): high-dose thoracic radiotherapy X-ray RT
  Interventions: Radiation: high-dose TRT
- standard-dose TRT (Active Comparator): standard-dose thoracic radiotherapy XRT
  Interventions: Radiation: standard-dose TRT

INTERVENTIONS:
Radiation: high-dose TRT — every day, Monday-Friday, for a total of 3 weeks, 45 Gy/ 3 Gy/ 15 f
  Arms: high-dose TRT
Radiation: standard-dose TRT — every day, Monday-Friday, for a total of 2 weeks, 30 Gy/ 3 Gy/ 10 f
  Arms: standard-dose TRT

SUMMARY:
Most patients with extensive stage small-cell lung cancer (ES-SCLC) who undergo chemotherapy, and prophylactic cranial irradiation, have persistent intrathoracic disease. A Dutch study recently proved that thoracic radiotherapy(TRT), using 30 Gy in 10 fractions of 3 Gy, could improve 2-year overall survival(OS) of this patient group compared with non-TRT group. But intrathoracic progression was still high, either with or without progression elsewhere, occurring in 43.7% in the TRT group. The ideal TRT regimen for ES-SCLC is undefined. Maybe higher dose can provide better local control(LC) and overall survival. In this study, the investigators propose to give an increased dose of TRT to determine whether higher dose will improve 2-year OS, LC and progression-free survival.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomised phase III study. For patients with ES-SCLC who respond to chemotherapy after four to six cycles of standard chemotherapy (platinum etoposide), 45Gy/15F of thoracic radiotherapy will be used in experimental arm, while 30Gy/10F of thoracic radiotherapy will be used in the control arm. Both survival and toxicity of the two arms will be observed and compared.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 70 years old, ECOG 0-2.
* Patients with histologically or cytologically proved small cell lung cancer.
* Extensive stage small-cell lung cancer (ES-SCLC), was characterized by tumors beyond the hemithorax, hilar, mediastinal, and supraclavicular nodes. According to 2007 AJCC cancer staging 7th edition, stage I-IIIB with lung metastases and stage IV should be defined as LD.
* Has 1-4 extracranial metastatic lesions.
* No brain or central nervous system (CNS) metastases.
* No prior history of anti-tumor treatment.
* Response after 4 to 6 cycles of EP-based chemotherapy within the past 4 weeks.
* No severe internal diseases and no organ dysfunction.
* Written informed consent provided.

Exclusion Criteria:

* Malignant tumors of other sites. Non melanoma skin cancer and Cervical carcinoma in situ were not included if curable.
* Active heart disease or acute myocardial infarction happen in six months.
* Psychiatric history.
* Pregnant woman or woman need to breast feed or woman with positive chorionic gonadotrophin (HCG).
* Uncontrolled diabetes or hypertension.
* Interstitial pneumonia or Active pulmonary fibrosis.
* Acute bacterial or fungal infection.
* Oral or intravenous use of steroids.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
overall survival | 2 years
  The time interval between diagnosis and death

SECONDARY OUTCOMES:
progression-free survival | 2 years
  The time interval between diagnosis and disease progression
Incidence of tumor recurrence in local or regional area | 2 years
  Number of patients experienceing recurrences in local or regional area divided by number of all enrolled patients
Incidence of radiotherapy and chemotherapy induced toxicities assessed by CTCAE v 4.0 | 2 years
  Number of patients experienceing any toxicities induced by radiotherapy or chemotherapy divided by number of all enrolled patients

CONTACTS AND LOCATIONS:
Overall Officials: LuHua Wang, MD, Principal Investigator — Cancer Hospital of CAMS
Locations (2):
- China (2):
  - Cancer Insititute and Hosiptal of Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Slotman BJ, van Tinteren H, Praag JO, Knegjens JL, El Sharouni SY, Hatton M, Keijser A, Faivre-Finn C, Senan S. Use of thoracic radiotherapy for extensive stage small-cell lung cancer: a phase 3 randomised controlled trial. Lancet. 2015 Jan 3;385(9962):36-42. doi: 10.1016/S0140-6736(14)61085-0. Epub 2014 Sep 14. PMID 25230595